CLINICAL TRIAL: NCT06623890
Title: An Observational, Multinational, Post-Marketing Registry of Omaveloxolone-Treated Patients With Friedreich's Ataxia
Brief Title: A Study to Learn More About the Long-Term Safety of BIIB141 (Omaveloxolone) in Participants With Friedreich's Ataxia Who Are Prescribed it by Their Own Doctors
Status: Recruiting | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 296FA401; EUPAS1000000196 (Other: HMA-EMA Catalogues)
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — omaveloxolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Omaveloxolone Naive Cohort: Participants with FA who will initiate omaveloxolone treatment per its approved label will be followed prospectively for up to 5 years.
  Interventions: Drug: Omaveloxolone
- Omaveloxolone Non-Naive Cohort: Participants with FA who initiated omaveloxolone treatment as per the approved label less than 12 months prior to enrollment in this study will be analyzed retrospectively (baseline data) followed by prospective analysis (post-baseline data) for up to 5 years.
  Interventions: Drug: Omaveloxolone

INTERVENTIONS:
Drug: Omaveloxolone — Administered as specified in the treatment arm.
  Other Names: SKYCLARYS; BIIB141

SUMMARY:
In this study, researchers will learn more about the safety of BIIB141, also known as omaveloxolone or SKYCLARYS®. This is a drug available for doctors to prescribe for people with Friedreich's Ataxia, also known as FA. This is known as an "observational" study, which collects health information about study participants without changing their medical care. Participants for this study will be found using a group called the Friedreich's Ataxia Global Clinical Consortium (FA GCC) UNIFIED Natural History Study (UNIFAI). The FA-GCC is a group of study research centers that helps provide clinical care for FA patients and also helps researchers learn more about how FA affects patients over a long time.

The main objective of this study is to collect safety information in participants with FA from UNIFAI. Some of the participants in this study will be prescribed BIIB141 for the first time by their own doctors. Some of the participants will have started taking BIIB141 after joining UNIFAI, but less than 12 months before joining this study.

The main questions researchers want to answer in this study are:

* How many participants had serious adverse events (SAEs)? An adverse event is considered serious when it results in death, is life-threatening, causes lasting problems, or requires hospital care.
* How many participants had adverse events (AEs) related to heart failure or liver damage caused by the drug?

Researchers will also learn more about :

• Why and when participants stopped treatment, left the study, or took more of the drug than was prescribed

This study will be done as follows:

* Participants will be screened to check if they can join the study.
* After joining the study, the participants who had never started BIIB141 treatment before must start it within 6 months. Otherwise, all participants will take BIIB141 throughout this study as prescribed by their own doctor.
* During the study, each participant's doctor will decide how often the participant visits the study research center to check on their health. This will be based on the doctor's own clinical judgment and what is recommended by the drug's label.
* Data from the participants' regular visits to their doctor will be collected at 1 month, 2 months, 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, and 60 months.
* Each participant will be in the study for up to 5 years.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the long-term safety of omaveloxolone as prescribed to participants with FA in the real-world setting, including characterization of all drug-induced liver injury (DILI) and congestive heart failure (CHF) AEs. The secondary objective of this study is to capture the reasons and timing of omaveloxolone treatment interruptions, discontinuations, and drug overdose.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented diagnosis of FA, including confirmation via genetic testing.
* Participants aged 16 years and older at initiation of omaveloxolone treatment.

For the omaveloxolone-naive cohort

- Initiating omaveloxolone treatment as per an approved label concurrent with enrolling in this study.

For the omaveloxolone-non-naive cohort

* Initiated omaveloxolone treatment as per an approved label less than 12 months prior to enrollment in this study
* Prior to enrollment, maintained omaveloxolone treatment with no discontinuation of more than 60 days
* Actively on treatment at the time of enrollment in this study
* Treating physician is the study site principal investigator or sub-investigator
* Study site confirms ability to provide required baseline data through medical record review, UNIFAI database, or other site-collected data
* Enrolled in the UNIFAI study prior to initiation of omaveloxolone treatment

Key Exclusion Criteria:

* Received off-label prescription of omaveloxolone at any time.
* Previously enrolled in a clinical trial of omaveloxolone.
* Participating in a blinded interventional trial at the time of enrollment in the study; participants may participate in other clinical trials after baseline data are collected.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants for this study will be identified and enrolled via the FA-Global Clinical Consortium (FA-GCC) UNIFIED Natural History Study (UNIFAI study).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Omaveloxolone Naive Cohort: Number of Participants With Treatment-Emergent Serious Adverse Events (TESAEs) | From the start of the treatment up to end of the study (up to 5 years)
Omaveloxolone Non-Naive Cohort: Number of Participants With Treatment-Emergent Serious Adverse Events (TESAEs) | From enrolment in the current study up to end of the study (up to 5 years)
Omaveloxolone Naive Cohort: Number of Participants With DILI and CHF AEs | From the start of the treatment up to end of the study (up to 5 years)
Omaveloxolone Non-Naive Cohort: Number of Participants With DILI and CHF AE | From enrolment in the current study up to end of the study (up to 5 years)

SECONDARY OUTCOMES:
Time to Omaveloxolone Treatment Interruption | Up to 5 years
Time to Omaveloxolone Treatment Discontinuation | Up to 5 years
Time to Omaveloxolone Drug Overdose | Up to 5 years
Number of Participants With Reasons for Omaveloxolone Treatment Interruption, Treatment Discontinuation and Overdose | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (14):
- United States (4):
  - UCLA Neurology, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Medizinische Universität Innsbruck, Innsbruck, Austria
- HUB-Hôpital Erasme, Brussels, Belgium
- Center for hereditary ataxias, Motol, Motol, Prague, Czechia
- Germany (3):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Würtemberg
  - University Hospital Aachen, Aachen
  - Klinikum der Universität München, Munich
- Italy (3):
  - Scientific Institute, IRCCS E. Medea, Conegliano
  - Fondazione I.R.C.C.S. Istituto Neurologico C. Besta, Milan
  - Ospedale Pediatrico Bambino Gesu, Rome
- Stichting Radboud universitair medisch centrum, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/